CLINICAL TRIAL: NCT01209455
Title: Mechanisms of N-acetylcysteine Mediated Vascular Adverse Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Gemma Watson, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NAC Forearm 0910
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Poisoning
Keywords: Acetylcysteine; Adverse effects; Acetaminophen; Anaphylactoid reactions
MeSH Terms: conditions — Poisoning; Anaphylaxis | interventions — Chlorpheniramine; Ranitidine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Saline (No Intervention): Volunteers will receive an incremental rising dose infusion of IA NAC (6 doses) together with a co-infusion of normal saline to determine a dose response curve for arterial vasodilatation in the forearm.
- Histamine antagonists (Active Comparator): Subjects will receive an increasing dose infusion of NAC as described in arm 1 but in this arm will receive a co-infusion of histamine antagonists (H1 and H2 antagonists) to determine vasodilatation in response to NAC in the presence of histamine antagonists.
  Interventions: Drug: Chlorphenamine and Ranitidine
- Low dose paracetamol (Active Comparator): Subjects will receive an increasing dose infusion of NAC as described in arm 1 but in this arm will receive a co-infusion of low dose paracetamol to determine whether the vasodilatory response to NAC is inhibited.
  Interventions: Drug: Paracetamol
- High dose paracetamol (Active Comparator): Subjects will receive an increasing dose infusion of NAC as described in arm 1 but in this arm will receive a co-infusion of higher dose paracetamol to determine whether the vasodilatory response to NAC is inhibited.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Chlorphenamine and Ranitidine — We intend to use chlorphenamine (H1 antagonist) and ranitidine (H2 antagonist).Assuming NAC causes vasodilatation with an increase in forearm blood flow, we propose to administer 5 mcg/min to ensure maximal H1 blockade. In the presence of increased forearm blood flow, we propose to administer 37.5 mcg/min.
  Arms: Histamine antagonists
Drug: Paracetamol — Therapeutic IV administration of 1g paracetamol results in a plasma concentration of ~12 mg/l. To achieve a desired concentration of ~25 mg/l, in the presence of a forearm blood blow of 50 ml/min, we would intend to administer an IA infusion of 1.25 mg/min. To account for the presence of increased forearm blood flow, we propose to administer 4 mg/min IA paracetamol.
  Arms: Low dose paracetamol
Drug: Paracetamol — To achieve a local paracetamol concentration of ~200 mg/l, a concentration comparable to potentially hepatotoxic concentrations following paracetamol overdose, we propose to administer 30 mg/min paracetamol.
  Arms: High dose paracetamol

SUMMARY:
Paracetamol overdose is the leading cause of acute liver failure in the Western World. N-acetylcysteine (NAC) has been the antidote of choice for over 30 years but its use is associated with adverse effects in 40% of cases. Patients characteristically experience nausea, vomiting and an anaphylactoid ('pseudo-allergic') syndrome. This reaction is clinically similar to true anaphylaxis (allergic reaction) including flushing, rash, constriction of airways, and a fall in blood pressure, but occurs via a different mechanism. Although treatable, these reactions lead to patient distress, commonly cause confusion among treating physicians, and lead to significant delays in antidote administration. The aetiology of these adverse reactions to NAC remains unclear. We hypothesise: i) these reactions result from a dose-dependent release of the chemical histamine, causing dilatation of blood vessels (vasodilatation) and the anaphylactoid syndrome; ii) paracetamol conversely exerts a protective effect on the reaction, with a less severe reaction observed in the presence of higher paracetamol concentrations. We will investigate the mechanisms underlying adverse reactions to NAC in the human forearm model, examining the role of histamine and other markers involved in the inflammatory process. The wider significance is an improved understanding of this poorly delineated phenomenon, with implications for other medications associated with similar reactions, such as non-steroidal anti-inflammatory drugs and opioids such as morphine.

DETAILED DESCRIPTION:
In this study the investigators test the following hypotheses:

1. NAC causes dose-dependent vasodilatation associated with histamine release in vivo.
2. Release of other mediators, known to be associated with anaphylaxis, does not occur during anaphylactoid reactions to NAC.
3. Paracetamol has a protective role against NAC adverse reactions.

Investigation of these hypotheses in man is difficult. While local skin changes to intradermal NAC have been used to examine dose-response in patients, this approach does not lend itself to detailed investigation of the underlying mechanism and cannot be used to explore the effect of high paracetamol concentrations. We propose to use an alternative well-established model previously used by us to investigate the mechanisms involved in the pharmacodynamics of morphine in man by the measurement of forearm blood flow and skin response following intra-arterial infusion. The proposed model allows administration of doses far smaller than those used systemically and thus minimises the risk of unwanted systemic effects from either NAC or paracetamol. Safe administration of intra-arterial NAC (up to 300 mg/min, greater than that intended here) has previously been demonstrated. Local changes can be used as a surrogate for systemic effects, as described previously.

We will take a structured 3-part approach to the research hypotheses. Studies 1 and 2 will aim to establish a dose-response curve and seek evidence of tachyphylaxis, while measuring the level of histamine release. The presence of tachyphylaxis may help to explain why, in the clinical setting, NAC can often be safely re-introduced following a reaction. In study 3, the investigators intend to conduct a 4-way randomised controlled crossover mechanistic study. This will examine the pharmacodynamic effect of NAC in both the presence and absence of histamine antagonists (antihistamines), and low- and high-dose paracetamol. This study will also enable investigation of a possible protective role of paracetamol.

For all studies, the investigators will recruit healthy male volunteers between the ages of 18 and 64 years. Subjects will be non-smokers on no concomitant medications. Individuals with clinically significant co-morbidity such as heart failure, hypertension, hyperlipidaemia, diabetes mellitus, asthma, coagulopathy or bleeding disorders will be excluded. Exclusion criteria will also include those individuals who have had recent infective or inflammatory conditions or recently donated blood (within the last 3 months).

Each study will be performed in a quiet, temperature-controlled room maintained at 22-24ºC with subjects lying supine. Participants will have fasted and abstained from caffeine and tobacco for at least 4 hours and from alcohol for 24 hours before each study.

Subjects will undergo cannulation of the brachial artery in one arm with a sterile 27-standard wire gauge steel needle. Study drugs will be infused via this cannula. Blood will be drawn from both the infused and control arms via 17-gauge venous cannulae inserted into each arm under local anaesthesia.

After a 30-min lead-in period, forearm blood flow will be measured at 6-10 minute intervals in the infused and non-infused arms by venous occlusion plethysmography using mercury-in-silastic strain gauges as described previously.

Subjects may be recruited to more than one study provided a minimum of 1 week has passed between studies.

Study 1: Dose-response study Sufficient volunteers will be recruited to complete 8 studies using an incremental rising dose infusion of intra-arterial NAC (6 doses) to determine a dose response curve for arterial vasodilatation in the forearm. After a washout period of 30 mins to ensure a return to normal state, this will be repeated to determine whether the response is consistent over time. Study 1 will identify a dose to be used in study 2 that causes maximum local forearm vasodilatation without systemic effects (rise in contralateral forearm blood flow, blood pressure, heart rate, facial flushing).

Our hypothesis is that while an increase in histamine may be observed in response to NAC, no change in the other mediators commonly associated with anaphylactic reactions will be demonstrated. Blood samples will be obtained at baseline, at the end of the study, and at 10-min intervals during the incremental dose infusion of NAC to include each of the 6 doses administered (total 14 occasions). To maximise efficiency in addressing our hypothesis we intend to measure histamine and NAC at each time point. Enough blood will also be drawn on each occasion for measurement of other potential inflammatory mediators, including tryptase, vWF, tPA, IL-6, PGD2, and PGI2.

Study 2: Acute tolerance study Acute tolerance will be investigated in study 2. Eight studies will be completed using a constant infusion of NAC over 60 mins at a dose identified in study 1. Forearm vasodilatation and the level of histamine release will be measured every 10 mins. This study may help to explain why in the clinical setting NAC can often be safely reintroduced, without complication, following a reaction.

Blood samples will be obtained at baseline, at the end of the study, and at 10-min intervals during the infusion of NAC (total 8 occasions). Histamine and NAC will be measured at each time point and blood stored for later measurement of other potential mediators if appropriate following the results of study 1.

Study 3: Mechanistic study

Study 3 is a 4-way randomised controlled crossover study to investigate potential mediators. Sufficient subjects will be recruited to complete 8 studies, with each volunteer attending 4 times. At each visit, subjects will receive an increasing dose infusion of NAC as described in study 1. In addition they will also receive one of:

1. Co-infusion of normal saline (control)
2. Co-infusion of histamine antagonists (H1 and H2 antagonist)
3. Co-infusion of low dose paracetamol to give a local concentration of <50 mg/l
4. Co-infusion of higher dose paracetamol to give a local concentration of ~200 mg/l

Blood samples will be obtained at baseline, at the end of the study, and at 10-min intervals during the incremental dose infusion of NAC to include each of the 6 doses administered (total 8 occasions). Histamine, NAC and paracetamol assays will be measured at all time points. Blood will also be stored for later analysis of the other mediators if appropriate according to the results of study 1.

Drugs We have previously administered intra-arterial NAC without complication. Assuming a forearm blood flow of 50 ml/min, an infusion of 25 mg/min would be expected to achieve a local concentration ~500 mg/l, similar to peak concentrations reached during the standard 20-hour intravenous NAC protocol used on the hospital wards. We intend to use a range of 6 incremental doses at 10 min intervals to include this concentration: 1 mg/min, 5 mg/min, 10 mg/min, 50 mg/min, 100 mg/min, and 200 mg/min. The total infusion rate will be maintained 1 ml/min.

Histamine antagonists in current clinical use have not yet been administered in intr-arterial studies. We intend to use chlorphenamine (H1 antagonist) and ranitidine (H2 antagonist). Intravenous (IV) administration of 10mg chlorphenamine results in a plasma concentration of ~14 mcg/l. IA administration of 1 mcg/min would achieve a similar forearm concentration. Assuming NAC causes vasodilatation with an increase in forearm blood flow, the investigators propose to administer 5 mcg/min to ensure maximal H1 blockade. Similarly, IV administration of 50mg ranitidine results in a plasma concentration of ~150 mcg/l. IA administration of 7.5 mcg/min would be expected to achieve a similar forearm concentration. In the presence of increased forearm blood flow, the investigators propose to administer 37.5 mcg/min.

Therapeutic IV administration of 1g paracetamol results in a plasma concentration of ~12 mg/l. To achieve a desired concentration of ~25 mg/l, in the presence of a forearm blood blow of 50 ml/min, the investigators would intend to administer an IA infusion of 1.25 mg/min. To account for the presence of increased forearm blood flow, the investigators propose to administer 4 mg/min IA paracetamol. To achieve a higher local PA concentration of ~200 mg/l, a concentration comparable to potentially hepatotoxic concentrations following PA overdose, the investigators propose to administer 30 mg/min PA.

Skin changes Skin changes will be assessed through assessment of erythema or oedema in the forearm recorded using the Modified Draize Scale. Subjects will also be asked to subjectively express the intensity of any itching on a scale of 1 (no itch) to 7 (intense itch).

Expertise available The studies will be carried out in the Clinical Research Facility at the Royal Infirmary of Edinburgh, which has extensive experience in performing such studies. Most of the assays will be undertaken in the University of Edinburgh laboratories, which have expertise in these assays. The principal investigator is a trainee clinical toxicologist with the necessary skills to undertake the research.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, non-smoking, volunteers aged between 18-64 years

Exclusion Criteria:

* Lack of informed consent Age <18 or >64 years Current smoker Current involvement in a clinical trial Clinically significant comorbidity: heart failure, hypertension, known hyper-lipidaemia, diabetes mellitus, asthma, coagulopathy or bleeding disorders Current intake of aspirin, other non-steroid anti-inflammatory medications, or vasodilators Recent infective/inflammatory condition Recent blood donation (during the preceding three months)

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-01-03 (Actual); Primary Completion 2011-07-15 (Actual); Study Completion 2011-07-15 (Actual)

PRIMARY OUTCOMES:
Attenuation of NAC induced vasodilatation by histamine antagonists (H1 and H2 antagonists) and/or paracetamol | 10, 20, 30, 40, 50, 60, 70, 80, 90 minutes

SECONDARY OUTCOMES:
Inhibition of the inflammatory cascade contributes to a paracetamol mediated protective role against NAC adverse reactions. | 10, 20, 30, 40, 50, 60, 70, 80, 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Euan A Sandilands, MRCP BSc, Principal Investigator — NHS Lothian
Locations (1):
- Clinical Research Facility, Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom